CLINICAL TRIAL: NCT06041542
Title: Evaluation of the Screening Effect of Artificial Intelligence Hand Activity Evaluation System for Cervical Spondylosis
Status: Completed | Type: Observational
Sponsor: Guangdong Provincial People's Hospital (Other)
Responsible Party: Principal Investigator, YunBing Chang, Head of spine Department, Guangdong Provincial People's Hospital
Other Study IDs: GDREC2020291H
Record Dates: First submitted 2022-07-03; First posted 2023-09-18 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: 10-second G&R Test
Keywords: 10-second G&R test; cervical spondylotic myelopathy; hand motion analysis; video analysis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Case group: Collect video of hand grasping from patients with cervical spondylotic myelopathy through intelligent video analysis system.
  Interventions: Diagnostic Test: 10-second hand grip and release test
- Control group: Collect video of hand grasping from normal people through intelligent video analysis system.
  Interventions: Diagnostic Test: 10-second hand grip and release test
- Differentiate group: Collect video of hand grasping from Stroke and Parkinson's disease through intelligent video analysis system.
  Interventions: Diagnostic Test: 10-second hand grip and release test

INTERVENTIONS:
Diagnostic Test: 10-second hand grip and release test — To grip and release hand in ten seconds

SUMMARY:
The purpose of this study:

1. Build an artificial intelligence screening tool for cervical spondylosis based on hand function analysis;
2. Verify the accuracy of cervical spondylosis screening tools.

DETAILED DESCRIPTION:
Cervical spondylotic myelopathy (CSM) has a high incidence in the middle-aged and elderly people. According to clinical research, the surgeon can makes a preliminary assessment of the severity of CSM based on a 10-second grip and release (G&R) test. The statistics of G&R test mainly rely on the surgeon's manual counting. When a patient's hand motion speed is too fast, the surgeon's manual counting is prone to error, leading to potential misdiagnosis. We construct and verify the intelligent video analysis system for Grip-&-release. The system has a high accuracy and inference speed that ensure the proposed model can be used as a screening examination tool for CSM and a medical assistance tool to help decision making during CSM treatment planning.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18-80 years old;
2. Patients who have received cervical CT or MR examination within the last month and have been clearly diagnosed or excluded from cervical spondylosis (i.e., those who have been clearly diagnosed before participating in the study);
3. People who are willing to participate in the study with CT/MR examination (i.e., those who have not been diagnosed before joining the study).

Exclusion Criteria:

1. Subjects with cervical spondylosis who have been examined but still cannot be definitively diagnosed or ruled out;
2. Subjects with definite presence of hand trauma;
3. People who do not have access to CT or MR;
4. Subjects who did not comply with the examination, were unable to perform neurological assessment, or were unable to fill out questionnaires.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1000 asymptomatic population in community; 200 cases of cervical spondylosis; Arthritis, Parkinson's disease, cerebral apoplexy 60 patients each.
Sampling Method: Non-Probability Sample
Enrollment: 1380 (Actual)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-12-30 (Actual)

PRIMARY OUTCOMES:
mJOA score | 2022-10-01-2022-12-30
  Correlate 10-second hand grip and release test with mJOA score

CONTACTS AND LOCATIONS:
Overall Officials: Yunbing Chang, M.D., Study Chair — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided